CLINICAL TRIAL: NCT02094352
Title: Randomized Controlled Trial of Subanesthetic Intravenous Ketamine Infusion in Conjunction With Continuous Epidural Infusion for Treatment of Refractory Complex Regional Pain Syndrome
Brief Title: Randomized Controlled Trial of Ketamine Infusion With Continuous Epidural Infusion for Treatment of Complex Regional Pain Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was unable to enroll efficiently despite trying various technique.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-003
Record Dates: First submitted 2013-12-23; First posted 2014-03-21 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Complex Regional Pain Syndrome
Keywords: Complex Regional Pain Syndrome; Pain management; Ketamine infusion
MeSH Terms: conditions — Complex Regional Pain Syndromes; Agnosia | interventions — Ketamine; Injections, Epidural; Control Groups; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine Infusion + Epidural Infusion + Booster Infusion (Experimental): Inpatient: Patients will receive a subanesthetic continuous intravenous infusion of KETAMINE 500mg/500ml in 0.9% Sodium Chloride with an epidural infusion.
  Outpatient: Patients will receive three ketamine booster infusions over the course of three months.
  Interventions: Drug: Ketamine Infusion + Epidural Infusion; Drug: Ketamine Booster Infusion
- Control Group + Epidural Infusion + Booster Infusion (Placebo Comparator): Inpatient: Patients will receive a subanesthetic continuous intravenous infusion of SALINE 500mg/500ml in 0.9% Sodium Chloride with an epidural infusion.
  Outpatient: Patients will receive three saline booster infusions over the course of three months.
  Interventions: Drug: Control Group + Epidural infusion; Drug: Control Group Booster Infusion

INTERVENTIONS:
Drug: Ketamine Infusion + Epidural Infusion — The ketamine and epidural infusions will be administered over 96 hours with appropriate titration.
  Other Names: Ketamine; Epidural
  Arms: Ketamine Infusion + Epidural Infusion + Booster Infusion
Drug: Control Group + Epidural infusion — The saline and epidural infusions will be administered over 96 hours with appropriate titration.
  Other Names: Epidural
  Arms: Control Group + Epidural Infusion + Booster Infusion
Drug: Ketamine Booster Infusion — Patients will receive three ketamine booster infusions over the course of three months.
  Other Names: Ketamine
  Arms: Ketamine Infusion + Epidural Infusion + Booster Infusion
Drug: Control Group Booster Infusion — Patients will receive three saline booster infusions over the course of three months.
  Other Names: Saline
  Arms: Control Group + Epidural Infusion + Booster Infusion

SUMMARY:
The purpose of this study is to determine whether epidural and ketamine infusions are effective in the treatment of Complex Regional Pain Syndrome (CRPS).

DETAILED DESCRIPTION:
Potential patients must clear all study requirements to be enrolled. Study requirements include labwork, psychiatric evaluation, and cardiology evaluation.

Once enrolled, patients will be in one of two groups:

1. Receives epidural infusion
2. Receives epidural and ketamine infusions

The patient and study staff are blinded.

This study requires multiple visits to Hospital for Special Surgery in New York City over the course of three months and concludes with a final visit after six months. The study will only cover costs associated with the scheduled in-patient and out-patient visits. The study patient will be responsible for all other costs (including travel and hotel accommodations) that he/she may incur for participating in this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must meet the Budapest CRPS criteria, including two or more symptom categories and three or more sign categories (as previously documented by a pain management physician or neurologist, or as observed on initial neurologic examination by the study investigator)
* Patients must have trialed at least three of the following therapies without relief judged adequate by the patient:
* Anti-depressants
* Anti-seizure medication
* Muscle relaxants
* Nerve blocks (somatic or sympathetic)
* Non-opioid analgesics
* Non-steroidal anti-inflammatory drugs
* Opioid analgesics
* Physical therapy
* Spinal cord stimulator trial
* Patients of either gender between the ages of 18 and 65 inclusive
* Patient report of a NRS pain score of at least 5 in at least two out-patient pain management physician clinic visits

EXCLUSION CRITERIA:

* Patients younger than 18 or older than 65
* Patients who:
* Are pregnant
* Are affected with glaucoma
* Are affected with thyrotoxicosis
* Are lactating
* Are on chronic anticoagulation therapy
* Have autonomic dysfunction with hemodynamic instability
* Have cardiac rhythm disturbance
* Have cerebrovascular disease
* Have conditions that would preclude central line placement
* Have conditions that would preclude epidural catheter placement
* Have congestive heart failure
* Have coronary artery disease
* Have creatinine level above 1.5
* Have electrolyte disturbance
* Have had previous reaction to IV contrast dye
* Have history of deep vein thrombosis
* Have history of systemic administration of ketamine for the treatment of pain
* Have liver disease
* Have known history of psychosis, significant thought disorder, or untreated (bipolar disorder depression or anxiety disorder ok)
* Have uncontrolled hypertension
* Any patient who is unable to provide consent due to cognitive difficulties
* Non-English speakers, as some of the instruments are only validated in English
* Patients with active litigation or workers compensation related to CRPS
* Patients with an intolerance or allergy to any medication planned as a component of the study
* Patients with known history of illegal drug use or alcohol dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2015-04-20 (Actual); Study Completion 2015-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Richman, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: Hospital for Special Surgery — http://www.hss.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Infusion + Epidural Infusion + Booster Infusion: Inpatient: Patients will receive a subanesthetic continuous intravenous infusion of KETAMINE 500mg/500ml in 0.9% Sodium Chloride with an epidural infusion.
  Outpatient: Patients will receive three ketamine booster infusions over the course of three months.
  Ketamine Infusion + Epidural Infusion: The ketamine and epidural infusions will be administered over 96 hours with appropriate titration.
  Ketamine Booster Infusion: Patients will receive three ketamine booster infusions over the course of three months.
- Control Group + Epidural Infusion + Booster Infusion: Inpatient: Patients will receive a subanesthetic continuous intravenous infusion of SALINE 500mg/500ml in 0.9% Sodium Chloride with an epidural infusion.
  Outpatient: Patients will receive three saline booster infusions over the course of three months.
  Control Group + Epidural infusion: The saline and epidural infusions will be administered over 96 hours with appropriate titration.
  Control Group Booster Infusion: Patients will receive three saline booster infusions over the course of three months.
Period: Overall Study
Arm/Group | Ketamine Infusion + Epidural Infusion + Booster Infusion | Control Group + Epidural Infusion + Booster Infusion
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Infusion + Epidural Infusion + Booster Infusion | Control Group + Epidural Infusion + Booster Infusion | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Reduction
Description: Evidence of changes in NRS pain scores between baseline and six months post infusion
Time Frame: 6 months post infusion
Population: Study terminated early due to lack of enrollment. We did not analyze any data.
Arm/Group | Ketamine Infusion + Epidural Infusion + Booster Infusion | Control Group + Epidural Infusion + Booster Infusion
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ketamine Infusion + Epidural Infusion + Booster Infusion | Control Group + Epidural Infusion + Booster Infusion
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes